CLINICAL TRIAL: NCT03534297
Title: A Phase 1b, Randomized, Double-Blinded, Dose Escalation, Single Center, Repeat-Dose Safety and Pharmacodynamics Study of Orally Administered Dapansutrile Capsules in Subjects With NYHA II-III Systolic Heart Failure
Brief Title: Study of Dapansutrile Capsules in Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Olatec Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OLT1177-06
Record Dates: First submitted 2017-12-21; First posted 2018-05-23 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Systolic Heart Failure
Keywords: heart failure; systolic heart failure
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure | interventions — dapansutrile

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to receive either dapansutrile capsules or placebo capsules in a 4:1 ratio within each Cohort.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a randomized, blinded, placebo-controlled study. Treatment allocation (to active or placebo treatment groups) will be blinded to all study participants, personnel, and investigators. Only the randomization statistician, drug labeling personnel and the medical monitor will be unblinded to the treatment assignment (in the event of an emergency, a scratch off label can be removed unmasking the treatment assignment to the PI and Medical Monitor).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- dapansutrile capsules (Experimental): A total of 8 patients in each cohort will receive dapansutrile capsules:
  * Cohort 1 will receive 5x 100 mg dapansutrile capsules QD for 14 days
  * Cohort 2 will receive 5x 100 mg dapansutrile capsules BID for 14 days
  * Cohort 3 will receive 5x 100 mg dapansutrile capsules QID for 14 days
  Interventions: Drug: dapansutrile capsules
- Placebo Capsules (Placebo Comparator): A total of 2 patients in each cohort will receive placebo capsules:
  * Cohort 1 will receive 5 placebo capsules QD for 14 days
  * Cohort 2 will receive 5 placebo capsules BID for 14 days
  * Cohort 3 will receive 5 placebo capsules QID for 14 days
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: dapansutrile capsules — Hard opaque capsules containing 100 mg of API.
  Other Names: OLT1177 capsules
  Arms: dapansutrile capsules
Drug: Placebo capsules — Hard opaque capsules containing 0 mg of API.
  Arms: Placebo Capsules

SUMMARY:
This is a Phase 1b randomized, double-blinded, single-center safety and pharmacodynamics study of sequential cohort, dose-escalating, repeat-dosing of dapansutrile or placebo (4:1 ratio) in subjects with stable systolic heart failure (HF) with LVEF≤40% symptomatic for NYHA functional classification II-III who show signs of systemic inflammation (high sensitivity plasma C reactive protein [hsCRP] > 2 mg/L). A total of 30 subjects will be enrolled in 3 sequential cohorts by randomized allocation (8 active and 2 placebo within each cohort). Progression to cohort 2 with dose escalation will occur following the Day 28 visit of the last subject in the first cohort. Progression to cohort 3 with dose escalation will occur following the Day 8 visit of the last subject in the second cohort.

Subjects will be screened and evaluated twice for eligibility: 1) at the time of Screening (up to 28 days prior to enrollment); and 2) at the Baseline visit, prior to randomization. Following enrollment, Baseline assessments will be conducted and the first dose of investigational product (either dapansutrile capsules or placebo capsules) will be administered at the clinical site upon completion of all assessment and collection of baseline parameters. Subjects will then self-administer investigational product once, twice or four times daily, depending on cohort, for up to fourteen (14) consecutive days beginning at the Baseline visit and continuing through the planned Day 14 visit. Subjects will return to the study clinic on Days 4, 8, 14 and 28 for follow-up visits. Additionally, subjects will be contacted for telephone follow-up on Day 42.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 years old or older
2. Symptomatic stable HF (NYHA class II-III) with reduced left ventricular ejection fraction (LVEF≤40%, measured within 6 months of enrollment - no changes in cardiac medications or new device implantation within past 2 months)
3. Peak exercise limited by shortness of breath and/or fatigue associated with a respiratory exchange ratio (RER) > 1.00 (reflecting maximal aerobic effort)
4. Reduced peak aerobic exercise capacity (peak VO2) to less than 80% of predicted value by age/gender at Baseline
5. Plasma CRP or hsCRP levels > 2 mg/L at Screening
6. Acceptable overall medical condition to be safely enrolled in and to complete the study (with specific regard to cardiovascular, renal and hepatic conditions) in the opinion of the Principal Investigator
7. Ability to provide written, informed consent prior to initiation of any study-related procedures, and ability, in the opinion of the Principal Investigator, to understand and comply with all the requirements of the study

Exclusion Criteria:

1. Women of childbearing potential, or men whose sexual partner(s) is a woman of childbearing potential who:

   1. Are or intend to become pregnant (including use of fertility drugs) during the study
   2. Are nursing
   3. Are not using an acceptable, highly effective method of contraception until all follow-up procedures are complete. (Acceptable, highly effective forms of contraception are defined as: oral contraception, intrauterine device, systemic [injectable or patch] contraception, double barrier methods, naturally or surgically sterile, strict abstinence or partner has been sterilized. If hormonal-based birth control is being used, subject or subject's sexual partner(s) must be on a stable-dose for ≥ 3 months prior to the Baseline visit and maintained at the same dosing level throughout the study.)
2. Abnormal blood pressure or heart rate response, angina or ECG changes (ischemia or arrhythmias) occurring during CPX
3. Presence or known history of autoimmune conditions (e.g., systemic lupus erythematosus, hypophysitis, etc.)
4. History or evidence of active tuberculosis (TB) infection at Baseline visit or one of the risk factors for tuberculosis such as but not limited or exclusive to:

   1. History of any of the following: residence in a congregate setting (e.g., jail or prison, homeless shelter, or chronic care facility), substance abuse (e.g., injection or non-injection), health-care workers with unprotected exposure to subjects who are at high risk of TB or subjects with TB disease before the identification and correct airborne precautions of the subject or
   2. Close contact (i.e., share the same air space in a household or other enclosed environment for a prolonged period (days or weeks, not minutes or hours)) with a person with active pulmonary TB disease within the last 12 months.
5. Use of any prohibited concomitant medications/therapies over the periods defined in Section 5.6.3 or planned use of any prohibited concomitant medications/therapies during the Treatment Period
6. Any other concomitant medical or psychiatric condition(s), disease(s) or prior surgery(ies) that, in the opinion of the Principal Investigator, would impair the subject from safely participating in the trial and/or completing protocol requirements, including but not limited to:

   1. physical inability to walk on a treadmill
   2. decompensated HF (edema, NYHA IV)
   3. significant ischemic heart disease, angina
   4. arterial hypotension (blood pressure [BP] systolic < 90 mmHg)
   5. arterial hypertension (resting BP systolic > 160 mmHg)
   6. atrial fibrillation with rapid ventricular response
   7. severe valvular disease
   8. severe chronic obstructive or restrictive pulmonary disease
   9. moderate-severe anemia (Hgb < 10 g/dL)
   10. severe diabetic neuropathy or myopathy
7. Active or recent (within 2 weeks) infection prior to the Baseline visit
8. History of or known positive for HIV, Hepatitis B surface antigen or antibodies to Hepatitis C Virus
9. Known history of renal impairment and/or creatinine clearance less than 50 mL/min calculated by Cockcroft-Gault method
10. Active malignancy or recent malignancy with chemotherapy treatment within the past 6 months
11. Enrollment in any trial and/or use of any investigational product or device within the immediate 30-day period prior to the Baseline visit
12. Previous exposure to the investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Adverse events | Screening through Day 42 follow-up
  Adverse events experienced by the patient will be recorded.

SECONDARY OUTCOMES:
Cardiopulmonary exercise test | Day 14
  Physician-supervised maximal aerobic exercise test will be administered using a metabolic cart that is interfaced with a motorized treadmill. Change in peak oxygen consumption in each group will be assessed.
Transthoracic Doppler ECG - Left Ventricle Ejection Fraction | Day 14
  Changes in left ventricular ejection fraction will be analyzed.
Transthoracic Doppler ECG - Left Ventricular Filling Pressure | Day 14
  Changes in estimated left ventricular filling pressure, measured as ratio of early diastolic transmitral pulsed wave Doppler flow velocity (E) to tissue Doppler velocity of the mitral annulus (e') will be analyzed.
Bioimpedance analysis | Day 14
  Bioimpedance is a non-invasive, quick and safe technique that allows to estimate body composition compartments (total body water, intracellular water, extracellular water, fat mass, fat-free mass, lean mass). Change in total body water will be assessed.
Kansas City Cardiomyopathy Questionnaire - Clinical Summary Score | Day 14
  Change in KCCQ score, a 23-item, self-administered instrument that independently measures a patient's perception of their health status, which includes heart failure symptoms. This scale is quantified in six domains: physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Each domain is scored on a 0-100 scale with 100 being better and 0 being worse. Two summary scores are calculated: the Clinical Summary Score (mean of symptom and physical function domain scores) and the Overall Summary Score (mean of the symptom, physical function, social limitations and quality of life scores).
Kansas City Cardiomyopathy Questionnaire - Overall Summary Score | Day 14
  Change in KCCQ score, a 23-item, self-administered instrument that independently measures a patient's perception of their health status, which includes heart failure symptoms. This scale is quantified in six domains: physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Each domain is scored on a 0-100 scale with 100 being better and 0 being worse. Two summary scores are calculated: the Clinical Summary Score (mean of symptom and physical function domain scores) and the Overall Summary Score (mean of the symptom, physical function, social limitations and quality of life scores).
Duke Activity Status Index | Day 14
  Change in Duke Activity Status Index, a self-administered questionnaire that measures a patient's functional capacity. The index consists of 12 "yes or no" questions, which are summed and used to calculate VO2peak and METS.
Vital signs - Pulse | Day 14
  Changes in pulse will be analyzed.
Vital signs - Blood Pressure | Day 14
  Changes in systolic and diastolic blood pressure will be analyzed.
Vital signs - Temperature | Day 14
  Changes in body temperature will be analyzed.
Vital signs - Respiratory Rate | Day 14
  Changes in respiratory rate will be analyzed.
Safety Laboratory Measurements - Chemistry | Day 14
  Changes in blood chemistry will be analyzed.
Safety Laboratory Measurements - Hematology | Day 14
  Changes in complete blood count will be analyzed.
Physical Examination | Day 14
  A full or targeted physical examination of the patient's major body systems
12-lead electrocardiogram | Day 8
  Electrodes will be placed on the patient to obtain a recording of the electrical activity of the heart.

OTHER OUTCOMES:
Pharmacokinetics | Baseline (pre and post dose), Day 4, Day 8, Day 14 and Day 28
  Blood sample for determination of dapansutrile blood concentrations.
Pharmacodynamics / Biomarkers | Baseline (pre and post dose), Day 4, Day 8, Day 14 and Day 28
  Blood sample for determination of levels of inflammatory biomarkers

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University - Pauley Heart Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Baat A, Trinh B, Ellingsgaard H, Donath MY. Physiological role of cytokines in the regulation of mammalian metabolism. Trends Immunol. 2023 Aug;44(8):613-627. doi: 10.1016/j.it.2023.06.002. Epub 2023 Jul 7. PMID 37423882
- [Derived] Wohlford GF, Van Tassell BW, Billingsley HE, Kadariya D, Canada JM, Carbone S, Mihalick VL, Bonaventura A, Vecchie A, Chiabrando JG, Bressi E, Thomas G, Ho AC, Marawan AA, Dell M, Trankle CR, Turlington J, Markley R, Abbate A. Phase 1B, Randomized, Double-Blinded, Dose Escalation, Single-Center, Repeat Dose Safety and Pharmacodynamics Study of the Oral NLRP3 Inhibitor Dapansutrile in Subjects With NYHA II-III Systolic Heart Failure. J Cardiovasc Pharmacol. 2020 Oct 24;77(1):49-60. doi: 10.1097/FJC.0000000000000931. PMID 33235030